CLINICAL TRIAL: NCT01192087
Title: Combined Treatment of Adenoid Cystic Carcinoma With Cetuximab and IMRT Plus C12 Heavy Ion Boost - ACCEPT - (ACC, Erbitux, and Particle Therapy); Phase I/II Feasibility Study
Brief Title: Adenoid Cystic Carcinoma, Erbitux, and Particle Therapy
Acronym: ACCEPT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Dept. of Radiation Oncology, INF 400, 69120 Heidelberg, Germany (Unknown); University Hospital Heidelberg (Other); Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Prof. Dr. Dr. J. Debus, Dept. of Radiation Oncology, INF 400, 69120 Heidelberg, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCEPT
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: adenoid cystic carcinoma; carbon ion therapy; IMRT (intensity-modulated therapy); radioimmunotherapy; Cetuximab
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab arm (Experimental): patients receive weekly cetuximab in combination with IMRT and carbon ion boost
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — cetuximab initial dose (7 days prior to RT treatment start): 400 mg/m² body surface cetuximab weekly doses (from RT treatment start throughout radiation treatment): 250 mg/m² body surface
  Other Names: Cetuximab (Erbitux)

SUMMARY:
The ACCEPT (A(denoid) c(ystic) c(arcinoma), E(rbitux, and) p(article) t(herapy))-trial is a prospective, monocentric phase I/II feasibility trial evaluating toxicity and efficacy in the combined treatment of intensity-modulated radiation therapy (IMRT) and carbon ion (C12) boost with the epidermal growth factor receptor (EGFR) antibody cetuximab. The primary objective of the study is to explore the toxicity of the combined modality regimen consisting of heavy ion therapy / IMRT and EGFR antibody immunotherapy, by assessing the rate of patients with mucositis or any other toxicity of severity grade 3 or 4 according to NCI CTCAE V. 4. Secondary endpoints include local control, distant control, overall disease-free survival, overall survival

DETAILED DESCRIPTION:
Treatment with novel radiotherapeutic technologies could increase local control in adenoid cystic carcinoma of the head and neck. Especially combined treatment with intensity-modulated radiation therapy and heavy ion (C12) boost to the primary tumor or previous tumor bed could be established as the treatment of choice in this disease.

Unfortunately, therapeutic results in the treatment of adenoid cystic carcinoma are still hampered by the occurrence of distant metastases (predominantly in the lungs) which, though progressing comparatively slowly, still limit the patient's life expectancy. Most adenoid cystic carcinomas (> 80%) though, exhibit over-expression of EGFR receptors and hence provide an approach for systemic treatment. In this prospective phase II trial, the application of the EGFR antibody cetuximab will be evaluated in combination with the established treatment of intensity-modulated radiation therapy plus C12 heavy ion boost.

The trial aims at evaluation of toxicity and feasibility of the combined treatment, as primary endpoint, as well as local control and disease-free survival as secondary endpoints.

ELIGIBILITY:
Inclusion criteria

* Histologically proven, or surgically resected adenoid-cystic carcinoma of the head and neck and
* macroscopic or microscopic residual tumor (R1/ R2) or
* Tumor stage >T3/T4 or
* perineural invasion and
* M0 stage
* Written informed consent
* Age between 18 and 70 years
* Karnofsky Index ≥ 70%
* Adequate bone-marrow, liver, and kidney function:
* neutrophils ≥ 1.5 x 109/L,
* thrombocytes ≥ 100 x 109/L,
* haemoglobin ≥ 10.0 g/dL
* bilirubin ≤ 2.0 g/dL
* SGOT, SGPT, AP, gamma-GT ≤ 3 x ULN
* serum creatinine ≤ 1.5 mg/dL
* effective contraception

Exclusion Criteria:

* Prior RT or chemotherapy for tumors of the head and neck
* R0 resection
* M1 (distant metastases)
* prior immunotherapy
* signs of active infection
* other serious illnesses
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction within the last twelve months, significant arrhythmias)
* Significant neurologic or psychiatric disorders including dementia or seizures
* Active disseminated intravascular coagulopathies
* Other serious underlying medical conditions prohibiting the patient's participation in the trial according to the judgement of the investigators
* Active participation in another clinical trial within the past 30 days
* Known allergic/ hypersensitivity reactions to non-human proteins
* Women: pregnant (Positive serum/ urine beta-HCG ) or breast-feeding,
* Known drug abuse,
* Other previous malignancy within the past 5 years, with exception of a history of a previous, adequately treated, basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix,
* Legal incapacity or limited legal capacity,
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with acute adverse effects as a Measure of toxicity | 6 weeks post completion of therapy
  The primary objective is to explore the toxicity of the combined treatment consisting of heavy ion therapy / IMRT and cetuximab by assessing the rate of patients with mucositis or any other toxicity of severity grade 3 or 4 according to NCI CTCAE V. 4.
  Acute treatment effects will be evaluated 6 weeks and late effects 3 years post completion of treatment
Number of Participants with late adverse effects as a Measure of toxicity | 3 years post completion of treatment
  The primary objective is to explore the toxicity of the combined treatment consisting of heavy ion therapy / IMRT and cetuximab by assessing the rate of patients with mucositis or any other toxicity of severity grade 3 or 4 according to NCI CTCAE V. 4.
  Acute treatment effects will be evaluated 6 weeks and late effects 3 years post completion of treatment

SECONDARY OUTCOMES:
local relapse-free survival | at 3 years post treatment
  Local relapse-free survival will be defined as the time from the initial dose of study therapy to the time of locoregional disease progression or relapse or death, or to the date of last assessment without any such event (censored observation)
distant relapse-free survival | at 3 years post treatment
  Distant relapse-free survival will be defined as the time from the initial dose of study therapy to the time of distant metastasis detection or death, or to the date of last assessment without any such event (censored observation)
overall disease-free survival | at 3 years post treatment
  Distant disease-free survival will be defined as the time from the initial dose of study therapy to the time of any detection of adenoid cystic carcinoma relapse or development of secondary cancer or death, or to the date of last assessment without any such event (censored observation)
overall survival | at 3 years post treatment
  The duration of survival will be determined by measuring the time interval from initial dose of study therapy to the date of death of any cause or last observation (censored)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Debus, Prof. Dr. Dr., Principal Investigator — Dept. of Radiation Oncology, INF 400, 69120 Heidelberg, Germany
Locations (1):
- Dept. of Radiation Oncology, Heidelberg, Germany

REFERENCES:
- [Background] Chen AM, Bucci MK, Weinberg V, Garcia J, Quivey JM, Schechter NR, Phillips TL, Fu KK, Eisele DW. Adenoid cystic carcinoma of the head and neck treated by surgery with or without postoperative radiation therapy: prognostic features of recurrence. Int J Radiat Oncol Biol Phys. 2006 Sep 1;66(1):152-9. doi: 10.1016/j.ijrobp.2006.04.014. PMID 16904520
- [Background] Munter MW, Schulz-Ertner D, Hof H, Nikoghosyan A, Jensen A, Nill S, Huber P, Debus J. Inverse planned stereotactic intensity modulated radiotherapy (IMRT) in the treatment of incompletely and completely resected adenoid cystic carcinomas of the head and neck: initial clinical results and toxicity of treatment. Radiat Oncol. 2006 Jun 6;1:17. doi: 10.1186/1748-717X-1-17. PMID 16756669
- [Background] Schulz-Ertner D, Nikoghosyan A, Didinger B, Munter M, Jakel O, Karger CP, Debus J. Therapy strategies for locally advanced adenoid cystic carcinomas using modern radiation therapy techniques. Cancer. 2005 Jul 15;104(2):338-44. doi: 10.1002/cncr.21158. PMID 15937907
- [Background] Schulz-Ertner D, Nikoghosyan A, Thilmann C, Haberer T, Jakel O, Karger C, Kraft G, Wannenmacher M, Debus J. Results of carbon ion radiotherapy in 152 patients. Int J Radiat Oncol Biol Phys. 2004 Feb 1;58(2):631-40. doi: 10.1016/j.ijrobp.2003.09.041. PMID 14751537
- [Background] Schulz-Ertner D, Nikoghosyan A, Jakel O, Haberer T, Kraft G, Scholz M, Wannenmacher M, Debus J. Feasibility and toxicity of combined photon and carbon ion radiotherapy for locally advanced adenoid cystic carcinomas. Int J Radiat Oncol Biol Phys. 2003 Jun 1;56(2):391-8. doi: 10.1016/s0360-3016(02)04511-x. PMID 12738314
- [Background] Jakel O, Kramer M, Schulz-Ertner D, Heeg P, Karger CP, Didinger B, Nikoghosyan A, Debus J. Treatment planning for carbon ion radiotherapy in Germany: review of clinical trials and treatment planning studies. Radiother Oncol. 2004 Dec;73 Suppl 2:S86-91. doi: 10.1016/s0167-8140(04)80022-7. PMID 15971317
- [Background] Huber PE, Debus J, Latz D, Zierhut D, Bischof M, Wannenmacher M, Engenhart-Cabillic R. Radiotherapy for advanced adenoid cystic carcinoma: neutrons, photons or mixed beam? Radiother Oncol. 2001 May;59(2):161-7. doi: 10.1016/s0167-8140(00)00273-5. PMID 11325445
- [Background] Douglas JG, Koh WJ, Austin-Seymour M, Laramore GE. Treatment of salivary gland neoplasms with fast neutron radiotherapy. Arch Otolaryngol Head Neck Surg. 2003 Sep;129(9):944-8. doi: 10.1001/archotol.129.9.944. PMID 12975266
- [Background] Pommier P, Liebsch NJ, Deschler DG, Lin DT, McIntyre JF, Barker FG 2nd, Adams JA, Lopes VV, Varvares M, Loeffler JS, Chan AW. Proton beam radiation therapy for skull base adenoid cystic carcinoma. Arch Otolaryngol Head Neck Surg. 2006 Nov;132(11):1242-9. doi: 10.1001/archotol.132.11.1242. PMID 17116822
- [Background] Mizoe JE, Tsujii H, Kamada T, Matsuoka Y, Tsuji H, Osaka Y, Hasegawa A, Yamamoto N, Ebihara S, Konno A; Organizing Committee for the Working Group for Head-And-Neck Cancer. Dose escalation study of carbon ion radiotherapy for locally advanced head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2004 Oct 1;60(2):358-64. doi: 10.1016/j.ijrobp.2004.02.067. PMID 15380567
- [Background] de Haan LD, De Mulder PH, Vermorken JB, Schornagel JH, Vermey A, Verweij J. Cisplatin-based chemotherapy in advanced adenoid cystic carcinoma of the head and neck. Head Neck. 1992 Jul-Aug;14(4):273-7. doi: 10.1002/hed.2880140403. PMID 1381339
- [Background] Kaplan MJ, Johns ME, Cantrell RW. Chemotherapy for salivary gland cancer. Otolaryngol Head Neck Surg. 1986 Sep;95(2):165-70. doi: 10.1177/019459988609500206. PMID 3035459
- [Background] Suen JY, Johns ME. Chemotherapy for salivary gland cancer. Laryngoscope. 1982 Mar;92(3):235-9. doi: 10.1288/00005537-198203000-00003. PMID 6279995
- [Background] Creagan ET, Woods JE, Rubin J, Schaid DJ. Cisplatin-based chemotherapy for neoplasms arising from salivary glands and contiguous structures in the head and neck. Cancer. 1988 Dec 1;62(11):2313-9. doi: 10.1002/1097-0142(19881201)62:113.0.co;2-4. PMID 3179947
- [Background] Dreyfuss AI, Clark JR, Fallon BG, Posner MR, Norris CM Jr, Miller D. Cyclophosphamide, doxorubicin, and cisplatin combination chemotherapy for advanced carcinomas of salivary gland origin. Cancer. 1987 Dec 15;60(12):2869-72. doi: 10.1002/1097-0142(19871215)60:123.0.co;2-y. PMID 2824016
- [Background] Venook AP, Tseng A Jr, Meyers FJ, Silverberg I, Boles R, Fu KK, Jacobs CD. Cisplatin, doxorubicin, and 5-fluorouracil chemotherapy for salivary gland malignancies: a pilot study of the Northern California Oncology Group. J Clin Oncol. 1987 Jun;5(6):951-5. doi: 10.1200/JCO.1987.5.6.951. PMID 3585449
- [Background] Laurie SA, Licitra L. Systemic therapy in the palliative management of advanced salivary gland cancers. J Clin Oncol. 2006 Jun 10;24(17):2673-8. doi: 10.1200/JCO.2005.05.3025. PMID 16763282
- [Background] Dodd RL, Slevin NJ. Salivary gland adenoid cystic carcinoma: a review of chemotherapy and molecular therapies. Oral Oncol. 2006 Sep;42(8):759-69. doi: 10.1016/j.oraloncology.2006.01.001. Epub 2006 Jun 6. PMID 16757203
- [Background] Airoldi M, Gabriele AM, Gabriele P, Pedani F, Marchionatti S, Succo G, Beatrice F, Bumma C. Concomitant chemoradiotherapy followed by adjuvant chemotherapy in parotid gland undifferentiated carcinoma. Tumori. 2001 Jan-Feb;87(1):14-7. doi: 10.1177/030089160108700103. PMID 11669550
- [Background] Haddad RI, Posner MR, Busse PM, Norris CM Jr, Goguen LA, Wirth LJ, Blinder R, Krane JF, Tishler RB. Chemoradiotherapy for adenoid cystic carcinoma: preliminary results of an organ sparing approach. Am J Clin Oncol. 2006 Apr;29(2):153-7. doi: 10.1097/01.coc.0000203756.36866.17. PMID 16601434
- [Background] Younes MN, Park YW, Yazici YD, Gu M, Santillan AA, Nong X, Kim S, Jasser SA, El-Naggar AK, Myers JN. Concomitant inhibition of epidermal growth factor and vascular endothelial growth factor receptor tyrosine kinases reduces growth and metastasis of human salivary adenoid cystic carcinoma in an orthotopic nude mouse model. Mol Cancer Ther. 2006 Nov;5(11):2696-705. doi: 10.1158/1535-7163.MCT-05-0228. PMID 17121916
- [Background] Vered M, Braunstein E, Buchner A. Immunohistochemical study of epidermal growth factor receptor in adenoid cystic carcinoma of salivary gland origin. Head Neck. 2002 Jul;24(7):632-6. doi: 10.1002/hed.10104. PMID 12112535
- [Background] Hotte SJ, Winquist EW, Lamont E, MacKenzie M, Vokes E, Chen EX, Brown S, Pond GR, Murgo A, Siu LL. Imatinib mesylate in patients with adenoid cystic cancers of the salivary glands expressing c-kit: a Princess Margaret Hospital phase II consortium study. J Clin Oncol. 2005 Jan 20;23(3):585-90. doi: 10.1200/JCO.2005.06.125. PMID 15659505
- [Background] Bonner JA, Harari PM, Giralt J, Azarnia N, Shin DM, Cohen RB, Jones CU, Sur R, Raben D, Jassem J, Ove R, Kies MS, Baselga J, Youssoufian H, Amellal N, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for squamous-cell carcinoma of the head and neck. N Engl J Med. 2006 Feb 9;354(6):567-78. doi: 10.1056/NEJMoa053422. PMID 16467544
- [Background] Alcedo JC, Fabrega JM, Arosemena JR, Urrutia A. Imatinib mesylate as treatment for adenoid cystic carcinoma of the salivary glands: report of two successfully treated cases. Head Neck. 2004 Sep;26(9):829-31. doi: 10.1002/hed.20094. PMID 15350030
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Derived] Adeberg S, Akbaba S, Lang K, Held T, Verma V, Nikoghosyan A, Bernhardt D, Munter M, Freier K, Plinkert P, Hauswald H, Herfarth K, Rieken S, Debus J, Jensen AD. The Phase 1/2 ACCEPT Trial: Concurrent Cetuximab and Intensity Modulated Radiation Therapy with Carbon Ion Boost for Adenoid Cystic Carcinoma of the Head and Neck. Int J Radiat Oncol Biol Phys. 2020 Jan 1;106(1):167-173. doi: 10.1016/j.ijrobp.2019.09.036. Epub 2019 Oct 3. PMID 31586664
- [Derived] Jensen AD, Nikoghosyan A, Hinke A, Debus J, Munter MW. Combined treatment of adenoid cystic carcinoma with cetuximab and IMRT plus C12 heavy ion boost: ACCEPT [ACC, Erbitux(R) and particle therapy]. BMC Cancer. 2011 Feb 15;11:70. doi: 10.1186/1471-2407-11-70. PMID 21320355